CLINICAL TRIAL: NCT03803371
Title: A PHASE IV, OPEN LABEL, RANDOMIZED, TWO TREATMENT, TWO PERIOD, TWO SEQUENCE, CROSSOVER BIOEQUIVALENCE STUDY TO COMPARE AN ORAL FORMULATION OF TRAMADOL HYDROCHLORIDE 37.5 MG/PARACETAMOL 325 MG TABLETS (TEST PRODUCT OF PFIZER) VERSUS ULTRACET(REGISTERED) (TRAMADOL HYDROCHLORIDE/PARACETAMOL 37.5 MG/325 MG OF JANSSEN CILAG FARMACÊUTICA LTDA, REFERENCE PRODUCT OF BRAZIL) IN HEALTHY ADULT RESEARCH SUBJECTS UNDER FASTING CONDITIONS
Brief Title: Bioequivalence Study of Tramadol Hydrochloride /Paracetamol Tablets Versus Ultracet Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B4741005
Record Dates: First submitted 2019-01-02; First posted 2019-01-14 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Healthy
MeSH Terms: interventions — Ultracet; Tramadol; Acetaminophen; Tablets; Drug Evaluation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tramadol hydrochloride 37.5 mg/Paracetamol 325 mg tablets (Experimental): Tramadol hydrochloride 37.5 mg/Paracetamol 325 mg tablets by mouth on Day 1 of period 1 or 2
  Interventions: Drug: Tramadol hydrochloride 37.5 mg/Paracetamol 325 mg tablets - tablet (Pfizer)
- Ultracet tablet (Active Comparator): Ultracet tablet (Tramadol hydrochloride 37.5 mg/Paracetamol 325 mg) by mouth on Day 1 of period 1 or 2
  Interventions: Drug: Ultracet Tablets

INTERVENTIONS:
Drug: Ultracet Tablets — Ultracet tablet (Janssen Cilag Farmacêutica Ltda) equivalent to Tramadol hydrochloride 37.5 mg/Paracetamol 325 mg
  Other Names: Reference drug
  Arms: Ultracet tablet
Drug: Tramadol hydrochloride 37.5 mg/Paracetamol 325 mg tablets - tablet (Pfizer) — Tramadol hydrochloride 37.5 mg/Paracetamol 325 mg tablets (Pfizer)
  Other Names: Test Drug
  Arms: Tramadol hydrochloride 37.5 mg/Paracetamol 325 mg tablets

SUMMARY:
The sponsor, Pfizer has developed a formulation of tramadol hydrochloride/ paracetamol 37.5 mg/ 325 mg (test drug) as a generic alternative to the reference listed product Ultracet®. In order to meet the requirements for registration as a generic drug, this study is being conducted to demonstrate the bioequivalence between the formulation of tramadol hydrochloride/ paracetamol 37.5 mg/ 325 mg provided by Pfizer and the reference drug tramadol hydrochloride/ paracetamol 37.5 mg/ 325 mg, available in the pharmaceutical market in Brazil (Ultracet®, Janssen Cilag Farmacêutica Ltda).

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy female research subjects and/or male research subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive.

Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:

1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause, and have a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
3. Have medically confirmed ovarian failure. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential.

   2. Body mass index (BMI) of 18.5 kg/m2 to 24.9 kg/m2 (the upper limit may vary up to 15% to allow subjects with a BMI from 18.5 kg/m2 to 28.6 kg/m2 to participate), and a total body weight >50 kg (>110 lbs).

   3. Evidence of a personally signed and dated informed consent document indicating that the research subject has been informed of all pertinent aspects of the study.

   4. Research subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures

   Exclusion Criteria:
   1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
   2. Clinically significant infections within the past 3 months (eg, those requiring hospitalization or parenteral antibiotics, or as judged by the Investigator), evidence of any infection within the past 7 days, history of disseminated herpes simplex infection or recurrent or disseminated herpes zoster.
   3. Any condition possibly affecting drug absorption (eg, gastrectomy, colon resection, etc.).
   4. Research subjects with a history of, or current evidence for, severe gastrointestinal narrowing (pathologic or iatrogenic).
   5. History of or current positive results for any of the following serological tests: hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), anti hepatitis C core antibody (HCV Ab), or human immunodeficiency virus (HIV) 1 and 2.
   6. Malignancy or a history of malignancy
   7. A positive urine drug test.
   8. A positive alcohol screen.
   9. History of regular alcohol consumption exceeding 14 drinks/week for female subjects or 21 drinks/week for male subjects [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor] within 6 months before screening.
   10. Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day.
   11. Treatment with an investigational drug within 6 months or 4 or 5 half lives preceding the first dose of investigational product (whichever is longer).
   12. Pregnant female subjects, breastfeeding female subjects, fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol from at least 14 days prior to the first dose of investigational product until at least 28 days after the last dose of investigational product.
   13. Use of prescription or nonprescription drugs and dietary supplements within 14 days or 5 half lives (whichever is longer) prior to the first dose of investigational product. Limited use of non prescription medications that are not believed to affect research subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.

       • Herbal supplements, hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone releasing intrauterine devices [IUDs], vaginal ring, and postcoital contraceptive methods), and hormone replacement therapy must have been discontinued at least 28 days prior to the first dose of investigational product.
   14. Consumption of grapefruit or grapefruit related citrus fruits (eg, Seville oranges, pomelos) or juices within 7 days prior to dosing.
   15. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 3 months prior to screening.
   16. History of sensitivity to heparin or heparin induced thrombocytopenia.
   17. History of hypersensitivity to tramadol or paracetamol or any of the components in the formulation of the study products.
   18. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
   19. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the research subject inappropriate for entry into this study.
   20. Research subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or research subjects who are the sponsor's employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Area under the tramadol and paracetamol plasma concentration-time curve from time zero to last time point (AUClast) | Predose (0 hour), at 0.08, 0.16, 0.25, 0.33, 0.41, 0.50, 0.66, 0.83, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12, 24 and 36 hours post dose
Maximum plasma concentrations of tramadol and paracetamol (Cmax) | Predose (0 hour), at 0.08, 0.16, 0.25, 0.33, 0.41, 0.50, 0.66, 0.83, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12, 24 and 36 hours post dose

SECONDARY OUTCOMES:
Area under the tramadol and paracetamol plasma concentration-time curve from time zero extrapolated to infinite time | Predose (0 hour), at 0.08, 0.16, 0.25, 0.33, 0.41, 0.50, 0.66, 0.83, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12, 24 and 36 hours post dose
Time to first occurrence of Cmax (Tmax) of tramadol and paracetamol | Predose (0 hour), at 0.08, 0.16, 0.25, 0.33, 0.41, 0.50, 0.66, 0.83, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12, 24 and 36 hours post dose
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Predose (0 hour), at 0.08, 0.16, 0.25, 0.33, 0.41, 0.50, 0.66, 0.83, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12, 24 and 36 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- ICF - Instituto de Ciencias Farmaceuticas de Estudos e Pesquisas Ltda, Aparecida de Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4741005&StudyName=A+PHASE+IV%2C+OPEN+LABEL%2C+RANDOMIZED%2C+TWO+TREATMENT%2C+TWO+PERIOD%2C+TWO+SEQUENCE%2C+CROSSOVER+BIOEQUIVALENCE+STUDY+TO+COMPARE+AN+ORAL+FORMULATION+OF+TRAMADOL+HYDROCHLORIDE+37.5+MG%2FPARACETAMOL+325+MG+TABLETS+%28TEST+PRODUCT+OF+PFIZER%29+VERSUS+ULTRACET%28REGISTERED%29+%28TRAMADOL+HYDROCHLORIDE%2FPARACETAMOL+37.5+MG%2F325+MG+OF+JANSSEN+CILAG+FARMAC%C3%8AUTICA+LTDA%2C+REFERENCE+PRODUCT+OF+BRAZIL%29+IN+HEALTHY+ADULT+RESEARCH+SUBJECTS+UNDER+FASTING+CONDITIONS